CLINICAL TRIAL: NCT04134507
Title: Multivariate Regression Analysis of Patient Satisfaction in Post-LASIK Patients With Presbyopia-Correcting IOLs vs. Post-LASIK Patients With Monofocal IOLs
Brief Title: Patient Satisfaction in Post-LASIK Patients With Presbyopia-Correcting IOLs vs. Post-Lasik Patients With Monofocal IOLs
Status: Completed | Type: Observational
Sponsor: Bucci Laser Vision Institute (Other)
Responsible Party: Sponsor
Other Study IDs: FAB-USA-001
Record Dates: First submitted 2019-10-17; First posted 2019-10-22 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Patient Satisfaction
Keywords: Post-LASIK; Presbyopia-correcting IOL; Monofocal IOL
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Extended Depth of Focus IOL: Post-LASIK patients with implantation of a presbyopia-correcting IOL
- Monofocal IOL: Post-LASIK patients with implantation of a monofocal IOL

SUMMARY:
Compare functional visual outcomes and patient satisfaction of post-LASIK patients having received presbyopia-correcting IOLs versus post-LASIK patients having received monofocal IOLs

ELIGIBILITY:
Inclusion Criteria:

* Post-LASIK
* Post cataract surgery
* Implantation of ZLB00, ZXR or ZXT, ZCB00, or AO60 intraocular lenses
* Spherical values greater than ± 0.50 and/or cylinder magnitude greater than 0.75D

Exclusion Criteria:

* Any vision-limiting problems (e.g., corneal, retinal, infection) which could potentially limit their post-operative visual potential
* Any newly acquired ocular condition or pathology (e.g., ARMD, epiretinal membrane, chronic dry eye, irregular astigmatism, diabetic retinopathy)
* Max sphere no greater than ± 0.50D and cylinder less than and/or equal to 0.75D

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Post-LASIK patients, male and female, aged 40 and older, who have undergone cataract surgery or clear lens exchange
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction: subjective questionnaire | Measured 3 months to 4 years after cataract surgery
  Subjective questionnaire explores the frequency and need for glasses for various visual functions at distance, intermediate, and near and overall satisfaction of visual function without glasses

SECONDARY OUTCOMES:
Visual Acuity at Distance | Measured 3 months to 4 years after cataract surgery
  Uncorrected and best corrected visual acuities measured at distance
Visual Acuity at Intermediate | Measured 3 months to 4 years after cataract surgery
  Uncorrected and best corrected visual acuities measured at intermediate
Visual Acuity at Near | Measured 3 months to 4 years; after cataract surgery
  Uncorrected and best corrected visual acuities measured at near

CONTACTS AND LOCATIONS:
Locations (1):
- Bucci Laser Vision, Wilkes-Barre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bucci FA Jr. Patient Satisfaction, Visual Outcomes, and Regression Analysis in Post-LASIK Patients Implanted With Multifocal, EDOF, or Monofocal IOLs. Eye Contact Lens. 2023 Apr 1;49(4):160-167. doi: 10.1097/ICL.0000000000000979. Epub 2023 Feb 22. PMID 36811831